CLINICAL TRIAL: NCT05842343
Title: Food Intake and IgA Microbiota in Anorexia Nervosa
Acronym: AAMIAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The coordinating investigator left the sponsor institution and has not been replaced.
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Laboratory Physiopathologie et biotherapies des infections muqueuses (GIMAP) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22CH356; 2023-A00318-37 (Other: ANSM)
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Anorexia Nervosa; Healthy Volunteer
Keywords: anorexia nervosa; microbiota; gut-brain-axis; immunology (IgA)
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acute anorexia nervosa (Experimental): patient diagnose for a first episode of pure restrictive anorexia nervosa will be included. They will have stool sample and Food intake evaluation.
  Interventions: Other: Stool sample; Other: Food intake evaluation
- Chronic anorexia nervosa (Experimental): Patient diagnose for anorexia nervosa at least 5 years ago and still maintaining a significant thinness will be included. They will have stool sample and Food intake evaluation.
  Interventions: Other: Stool sample; Other: Food intake evaluation
- Healthy control (Placebo Comparator): Healthy Patient will be included. They will have stool sample and Food intake evaluation.
  Interventions: Other: Stool sample; Other: Food intake evaluation

INTERVENTIONS:
Other: Stool sample — Purification by affinity of the IgA coated bacteria from a fecal solution. Genomic analysis of the bacteria for diversity and richness
Other: Food intake evaluation — Measure (by survey) of food group intake for : lipids /proteins / fibers / carbohydrates

SUMMARY:
Anorexia nervosa is characterized by intestinal dysbiosis, related to the feeding behavior impairment presented by these patients. Pathophysiologic hypotheses are involving the trouble of the microbiota-gut-brain axis in the field of mental diseases.

DETAILED DESCRIPTION:
Anorexia nervosa is characterized by intestinal dysbiosis, related to the feeding behavior impairment presented by these patients. Here we aim to characterize the IgA-coated fraction of bacteria from the intestinal microbiota, linked to the regulation of the mucosal immune system and the epithelium physiology. Abnormalities of this microbiota are reported in inflammatory bowel disease and are associated to immune trouble. As food intake plays a key role in shaping microbiota, we aim to correlate data from IgA microbiota to food intake specificity, and to anorexia nervosa phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* female subject, adult, affiliated to a social security system, under the care of the eating disorder department of university hospital of st Etienne
* presenting a diagnosis of pure restrictive anorexia nervosa.

For acute subgroup : BMI between 11 and 17.5 kg/m2, patient with a first episode of restrictive anorexia nervosa or with hyperphagic episodes.

For the chronic subgroup: BMI between 11 and 17.5 kg/m2, disease evolving for more than 5 years.

For Healthy volunteer: BMI between 20 and 24 kg/m², stable weight for the last 3 months, no eating disorder or history of eating disorder

Exclusion Criteria:

* patient does not understand French.
* laxative treatment in progress or stopped for less than 15 days,
* antibiotic treatment in the two months preceding inclusion,
* pre-pro or symbiotic treatment in progress or in the month preceding inclusion,
* patient with one of the following comorbid disorders: celiac disease, chronic inflammatory bowel disease, lactose intolerance, unstabilized hyperthyroidism, unstabilized diabetes,
* subject under legal protective measures.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Total microbiotic profile | 1 week after inclusion
  abundance and diversity parameters of the IgA microbiota fraction of the intestinal microbiota obtained by 16s rDNA analysis of stool suspension samples from acute anorexia nervosa, chronic anorexia nervosa and control subjects.

SECONDARY OUTCOMES:
ELISA assay of fecal immunoglobulins | 1 week after inclusion
  ELISA determination of immunoglobulin A and immunoglobulin M in the stool of acute anorexia nervosa, chronic anorexia nervosa and control subjects.
Microbiotic profile of total intestinal microbiota | 1 week after inclusion
  Total microbiotic profile (abundance and diversity) of the intestinal microbiota obtained by 16s rDNA analysis of stool suspension samples from acute anorexia nervosa, chronic anorexia nervosa and control subjects.
Food intake characteristics | 1 week after inclusion
  Qualitative and quantitative assessment of dietary intake by a dietary survey of acute anorexia nervosa, chronic anorexia nervosa and control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan GABRIEL-SEGARD, Md, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No